CLINICAL TRIAL: NCT01303822
Title: Mindfulness-based Stress Reduction in Supportive Cancer Treatment: Effects of a Day-care Clinic Group Program on Psychometric Parameters in Cancer Patients (Stressbewältigung Durch Achtsamkeit in Der Supportiven Onkologischen Therapie (SASO): Auswirkung Eines Tagesklinischen Gruppenprogramms Auf Psychometrische Parameter Bei Krebspatienten)
Brief Title: Mindfulness-based Stress Reduction in Cancer Treatment
Acronym: SASO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Holger Cramer, Research fellow, Universität Duisburg-Essen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-4600
Record Dates: First submitted 2011-02-24; First posted 2011-02-25 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2013-07

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mindfulness-based day-care clinic group program (Experimental): 11 weeks of mindfulness-based day-care clinic group program. 6 hours per week.
  Interventions: Behavioral: Mindfulness-based day-care clinic group program

INTERVENTIONS:
Behavioral: Mindfulness-based day-care clinic group program — 11 weeks of mindfulness-based day-care clinic group program. 6 hours per week.

SUMMARY:
Emotional and mental symptoms are common consequences of cancer diagnosis and treatment. Coping with these symptoms seems to be influenced by interpretation of illness, locus of health control and spiritual attitudes in dealing with illness.

Mindfulness-based stress reduction has been shown to reduce physical and mental symptoms in cancer patients.

The aim of this study is to investigate the effect of a mindfulness-based day-care clinic group program on quality of life, anxiety and depression in cancer patients and to evaluate the association with coping styles, spiritual attitudes in dealing with illness, mindfulness and interpretation of illness.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cancer
* Physical and mental ability to participate in the program

Exclusion Criteria:

* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2011-03; Primary Completion 2013-03 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life | Week 11
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30).
  Reference: Carlson LE, Speca M, Patel KD, Goodey E. Mindfulness-based stress reduction in relation to quality of life, mood, symptoms of stress, and immune parameters in breast and prostate cancer outpatients. Psychosom Med. 2003;65:571-581.

SECONDARY OUTCOMES:
Health-related quality of life | Week 32
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30).
  Reference: Carlson LE, Speca M, Patel KD, Goodey E. Mindfulness-based stress reduction in relation to quality of life, mood, symptoms of stress, and immune parameters in breast and prostate cancer outpatients. Psychosom Med. 2003;65:571-581.
Anxiety and depression | Week 11; week 32
  Hospital Anxiety and Depression Score (HADS)
Life satisfaction | Week 11; week 32
  Brief Multidimensional Life Satisfaction Scale (BMLSS).
  Reference: Büssing A, Fischer J. Interpretation of illness in cancer survivors is associated with healthrelated variables and adaptive coping styles. BMC Womens Health. 2009;9:2.
Mindfulness | Week 11; week 32
  Freiburg Mindfulness Inventory (FMI). Reference:Walach H, Buchheld N, Buttenmüller V, Kleinknecht N, Grossmann P, Schmidt S (2003). Empirische Erfassung der Achtsamkeit - Die Konstruktion des Freiburger Fragebogen zur Achtsamkeit (FFA) und weitere Validierungsstudien. In Heidenreich T, Michalak J: Achtsamkeit und Akzeptanz in der Psychotherapie, dgvt-Verlag.
Adaptive coping styles | Week 11; week 32
  AKU questionnaire.
  Reference: Büssing A, Fischer J. Interpretation of illness in cancer survivors is associated with healthrelated variables and adaptive coping styles. BMC Womens Health. 2009;9:2.
Spiritual and religious attitudes in dealing with illness | Week 11; week 32
  SpREUK questionnaire.
  Reference: Büssing A. Spirituality as a resource to rely on in chronic illness: the SpREUK questionnaire. Religions 2010;1:9-17.
Interpretation of illness | Week 11; week 32
  Interpretation of Illness Questionnaires (IIQ).
  Reference: Büssing A, Fischer J. Interpretation of illness in cancer survivors is associated with healthrelated variables and adaptive coping styles. BMC Womens Health. 2009;9:2.

CONTACTS AND LOCATIONS:
Locations (1):
- Kliniken Essen-Mitte, Knappschafts-Krankenhaus, Department for Internal and Integrative Medicine, Essen, North Rhine-Westphalia, Germany